CLINICAL TRIAL: NCT01957358
Title: Resolving Grief and Moving On After Spinal Cord Injury
Brief Title: Resolving Grief After Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Karen Ethans (Other)
Responsible Party: Sponsor-Investigator, Dr. Karen Ethans, Director, Spinal Cord Injury Rehabilitation Program, University of Manitoba
Organization: University of Manitoba (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: GR2013
Record Dates: First submitted 2013-09-26; First posted 2013-10-08 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle counselling using the Grief Recovery Method (Experimental): Volunteers will participate in a series of weekly and twice-weekly sessions with a counselor who has obtained special training in the Grief Recovery Method.
  Interventions: Behavioral: The Grief Recovery Method

INTERVENTIONS:
Behavioral: The Grief Recovery Method — The Grief Recovery Method is a structured process designed to help people with spinal cord injuries examine their knowledge of their injury, their emotional reaction to their injury, and their ability to acknowledge their grief over the injury in order to learn techniques to resolve the grief in order to achieve a more complete recovery. Participants will attend a total of 18 sessions, some one-on-one, and some in a group setting. The Grief Recovery Handbook, handouts, DVD (digital video disc) presentations and questionnaires will be used. Targeted activities to decrease isolation and assist volunteers to identify goals for recovery will be utilized.

SUMMARY:
The purpose of this study is to examine the usefulness of the Grief Recovery Method in assisting persons with spinal cord injuries to achieve as complete a recovery as possible, thereby allowing for fuller participation in life.

ELIGIBILITY:
Inclusion Criteria:

* Persons with a spinal cord injury who are willing to participate in the program.

Exclusion Criteria:

* Unable or unwilling to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2013-10; Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Impact of Event Scale | At Sessions 1 and 18. (Baseline and month 4)
  A self-administered questionnaire with 22 questions designed to measure the subjective response to a specific traumatic event (for this study, the event is the spinal cord injury).

SECONDARY OUTCOMES:
Modified Grief Inventory | At Sessions 1and 18 (baseline and month 4).
  A self-reported 2-part questionnaire that asks the volunteer to circle responses to questions about past behavior and present feelings about their spinal cord injury.
The Coping with Health Injuries and Problems | At sessions 1 and 18 (Baseline and month 4)
  A 32-question self-reported scale that measures coping with illness.

CONTACTS AND LOCATIONS:
Locations (1):
- WRHA Health Sciences Centre Rehabilitation Hospital, Winnipeg, Manitoba, Canada